CLINICAL TRIAL: NCT04243655
Title: Use of HA 330-II for Hemofiltration in Patients With Acute Liver Failure as a Bridge to Liver Transplantation: Clinical Evaluation Protocol.
Brief Title: Use of HA 330-II for Hemofiltration in Patients With ALF as a Bridge to Liver Transplantation .
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIG-G/ALFLD
Record Dates: First submitted 2020-01-17; First posted 2020-01-28 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Acute-On-Chronic Liver Failure
MeSH Terms: conditions — Acute-On-Chronic Liver Failure

STUDY DESIGN:
Intervention Model Description: Hemoperfusion treatment with HA 330-II, one unit for 2-4 hours treatment, for 3 consecutive days along with standard medical treatment (SMT) as per patients requirement.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hemoperfusion treatment with HA 330-II (Experimental): Hemoperfusion treatment with HA 330-II, one unit for 2-4 hours treatment, for 3 consecutive days along with SMT as per patients requirement.
  Interventions: Device: HA 330-II; Drug: Standard medical treatment (SMT)
- Standard medical treatment (SMT) (Active Comparator): SMT as per patients requirement- Management of cerebral edema/intracranial hypertension: prophylactic antibiotics, administration of mannitol or 3% saline for severe elevation of Intra Cranial Pressure, volume replacement and pressor support (noradrenaline, doubutamine, dopamine) as needed, NAC and correction of metabolic parameters.
  Interventions: Drug: Standard medical treatment (SMT)

INTERVENTIONS:
Device: HA 330-II — One unit for 2-4 hours treatment, for 3 consecutive days
  Arms: Hemoperfusion treatment with HA 330-II
Drug: Standard medical treatment (SMT) — SMT as per patients requirement- Management of cerebral edema/intracranial hypertension: prophylactic antibiotics, administration of mannitol or 3% saline for severe elevation of Intra Cranial Pressure, volume replacement and pressor support (noradrenaline, doubutamine, dopamine) as needed, NAC and correction of metabolic parameters.

SUMMARY:
ALF (ALF) is defined by three criteria: (1) rapid development of hepatocellular dysfunction (jaundice, coagulopathy), (2) hepatic encephalopathy, and (3) absence of a prior history of liver disease.

Interval between onset of acute hepatic injury (jaundice) and onset of liver failure (encephalopathy with or without coagulopathy) in such patients (icterus-encephalopathy interval; IEI) has been described to be between 4 weeks (Indian definition) to 24 weeks (AASLD-ALF study group). Further, due to the diverse natural course, ALF has been sub-classified as hyperacute (IEI ≤ 7 day), acute (IEI ≤ 4 weeks) and sub-acute ALF (IEI ≥ 5 week to ≤12 weeks) by British authors.

DETAILED DESCRIPTION:
Since the 1960s, Liver Transplantation (LT) has emerged as a cornerstone intervention to cure liver failure. Mortality in patients with liver failure who cannot be rescued with Liver Transplantation remains high despite improvements in supportive care.

Artificial Liver Support System (ALSS) in ALF aim to remove excess inflammatory cytokines and attenuate inflammatory response, to remove albumin-bound and water-soluble toxins, to restore and preserve hepatic function and mitigate or limit the progression of multiorgan failure while hepatic recovery or liver transplant occurs. ALSS may also provide benefit in instances where LT is contraindicated.

The following beneficial effects have been documented with ALSS in ALF patients: improvement of jaundice, amelioration of hemodynamic instability, improvement of hepatic encephalopathy, SOFA score and survival.

HA 330-II is a broad-spectrum adsorbent made of neutral macroporous resin, removes toxins such as Inflammatory mediators (IL-1, IL-6, IL-8 & TNF-α) along with hepatic toxins such as phenol, mercaptan, aromatic amino acids, false neurotransmitters and indirectly ammonia by improving liver function recovery. However, this indirect ammonia removal with HA 330-II is insignificant. By removing excess inflammatory cytokines and attenuating uncontrolled immune response, HA 330-II prevents worsening of encephalopathy, improves liver function recovery and improves prognosis.

ELIGIBILITY:
Inclusion Criteria:

• Acute Liver Failure patients with SIRS and Hepatic Encephalopathy, without hyperbilirubinemia.

Exclusion Criteria:

* Patients with age less than 18 years or more than 65 years
* Extremely moribund patients with an expected life expectancy of less than 24 hours or with poor prognosis
* With poor blood clotting function and PTA <30%.
* Active Bleed
* Chronic heart, lung or kidney disease
* Malignant tumors including liver cancer
* Past history of organ transplantation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-12-30 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy of HA 330-II to prolong liver-transplantation free survival. | Up to 30 Days
  The length of survival time after first hemofiltration treatment during the follow-up period.

SECONDARY OUTCOMES:
Change in Systemic inflammatory response syndrome (SIRS) score. | Up to 7 Days, post hemofiltration
  To assess efficacy of treatment.
Change in Acute Physiology and Chronic Health Evaluation (APACHE-II) score. | Up to 7 Days, post hemofiltration
  To assess efficacy of treatment.
Change in sequential organ failure assessment (SOFA) score. | Up to 7 Days, post hemofiltration
  To assess efficacy of treatment.
Change in chronic liver failure-sequential organ failure assessment (CLIF-SOFA) score. | Up to 7 Days, post hemofiltration
  To assess efficacy of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Mithun Sharma, Principal Investigator — AIG Hospitals
Locations (1):
- Asian Institute Of Gastroenterology, Hyderabad, Telangana, India

REFERENCES:
- [Background] Rolando N, Wade J, Davalos M, Wendon J, Philpott-Howard J, Williams R. The systemic inflammatory response syndrome in acute liver failure. Hepatology. 2000 Oct;32(4 Pt 1):734-9. doi: 10.1053/jhep.2000.17687. PMID 11003617
- [Background] Lee KC, Stadlbauer V, Jalan R. Extracorporeal liver support devices for listed patients. Liver Transpl. 2016 Jun;22(6):839-48. doi: 10.1002/lt.24396. PMID 26785141
- [Background] Larsen FS, Schmidt LE, Bernsmeier C, Rasmussen A, Isoniemi H, Patel VC, Triantafyllou E, Bernal W, Auzinger G, Shawcross D, Eefsen M, Bjerring PN, Clemmesen JO, Hockerstedt K, Frederiksen HJ, Hansen BA, Antoniades CG, Wendon J. High-volume plasma exchange in patients with acute liver failure: An open randomised controlled trial. J Hepatol. 2016 Jan;64(1):69-78. doi: 10.1016/j.jhep.2015.08.018. Epub 2015 Aug 29. PMID 26325537